CLINICAL TRIAL: NCT00781599
Title: Improving Medication Compliance and Smoking Cessation Treatment Outcomes for African American Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nikki Nollen, PhD, MA (Other)
Responsible Party: Sponsor-Investigator, Nikki Nollen, PhD, MA, Assistant Professor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11500
Record Dates: First submitted 2008-10-27; First posted 2008-10-29 (Estimated); Results first posted 2012-06-27 (Estimated); Last update posted 2012-07-11 (Estimated); Status verified 2012-06

CONDITIONS: Smokers
Keywords: African american; smokers; smoking cessation; African American smokers
MeSH Terms: conditions — Smoking Cessation | interventions — Varenicline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Chantix for 3 months and Standard Counseling
  Interventions: Drug: Chantix; Behavioral: Standard Counseling
- 2 (Experimental): Chantix for 3 months and Adherence Counseling
  Interventions: Drug: Chantix; Behavioral: Adherence Counseling; Behavioral: Standard Counseling

INTERVENTIONS:
Drug: Chantix — Chantix 0.5 mg once daily on days 1-3, 0.5 mg twice daily on days 4-7, and 1 mg twice daily on day 8 through end of treatment at month 3
  Other Names: varenicline
Behavioral: Adherence Counseling — Induction Support counseling on days 8, 12, 20 and months 1 and 2. Adherence counseling based on the Information-Motivation-Behavioral Skills model of adherence behavioral change.
  Arms: 2
Behavioral: Standard Counseling — Visit with counselor on Day 8 to develop a plan to quit smoking. Discuss strategies to quit, risks of continued smoking and discuss strategies for coping with withdrawal and craving.

SUMMARY:
Little is known about the support needed to improve compliance with Chantix for smoking cessation. This is a two arm pilot study of African American smokers to provide varying levels of side effect management and compliance support during a 12 week treatment period. The primary aim of the study is to estimate the effect of induction support compared to standard care in increasing compliance with Chantix at month 3

ELIGIBILITY:
Inclusion Criteria:

* African American
* 18-75 years of age
* Smoke more than 10 cigarettes per day
* Have a functioning telephone number
* Be interested in quitting smoking
* Be willing to take 3 months of Chantix
* Be willing to complete all study visits

Exclusion Criteria:

* Renal impairment
* Evidence or history of clinically significant allergic reactions to Chantix
* Cardiovascular event in the past month
* History of alcohol or drug abuse/dependency in the past year
* Major depressive disorder in the last year requiring treatment
* History of panic disorder
* Psychosis, bipolar or eating disorder
* Use of antidepressants, antipsychotics, mood stabilizers/anticonvulsants or naltrexone
* Use of tobacco products other than cigarettes
* Use of nicotine replacement therapy, bupropion, clonidine or nortriptyline in the month prior to enrollment
* Prior use of Chantix
* Women who are pregnant, contemplating getting pregnant or breastfeeding
* Plans to move from Kansas City during the 3 month treatment phase
* Another household member enrolled in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2008-10; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Nollen, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

REFERENCES:
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were randomized between March and August 2009. Participants were recruited from Swope Health Central.
Groups:
- Chantix for 3 Months, Standard Counseling: Participants received Chantix for 3 months. Participants received verbal instructions on how to take the medication. Participants met with a study counselor during randomization visit to develop a plan to quit.
- Chantix for 3 Months and Adherence Counseling: Participants received Chantix for 3 months. Participants received verbal instructions on how to take the medication. Participants met with a study counselor during randomization visit to develop a plan to quit. Participants received 5 additional counseling sessions. Adherence counseling based on the Information-Motivation-Behavioral Skills model.
Period: Overall Study
Arm/Group | Chantix for 3 Months, Standard Counseling | Chantix for 3 Months and Adherence Counseling
Started | 36 | 36
Completed | 29 | 32
Not Completed | 7 | 4
Not completed — Lost to Follow-up | 7 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chantix for 3 Months, Standard Counseling | Chantix for 3 Months and Adherence Counseling | Total
Number analyzed (Participants) | 36 | 36 | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 36 | 34 | 70
  >=65 years | 0 | 2 | 2
Age Continuous [Mean (Standard Deviation); unit: years] | 44.3786 (11.046) | 49.1980 (11.222) | 46.788 (11.320)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 12 | 33
  Male | 15 | 24 | 39
Region of Enrollment [Number; unit: participants]
  United States | 36 | 36 | 72

OUTCOME MEASURES:

1. Primary Outcome: Percent Compliance With Chantix
Description: Compliance with Chantix calculated as the total doses taken over the total number of doses prescribed. Adherence was measured by pill counts. Measurements taken during monthly medication refill visits. There was no specific predetermined cutoff number on the scale which determined non-compliance. All results from compliance calculations are included in the table.
Time Frame: Months 1, 2, 3
Population: Number of participants determined by total number of enrolled participants. For reporting purposes, those participants that did not show up for a visit were treated as smokers.
Measure: Mean (Standard Deviation); unit: Percentage of Participants
Arm/Group | Chantix for 3 Months, Standard Counseling | Chantix for 3 Months and Adherence Counseling
Number analyzed (Participants) | 36 | 36
Percentage of Participants
  Month 1 | 90.7 (9.5) | 85.8 (23.0)
  Month 2 | 87.1 (18.9) | 91.7 (17.4)
  Month 3 | 89.2 (24.4) | 82.1 (36.4)

2. Secondary Outcome: Cotinine Verified 7 Day Point Prevalence Smoking Abstinence
Description: Smoking cessation verified by salivary cotinine (COT). A COT of <20 ng/ml indicated smoking abstinence.
Time Frame: Month 3
Population: A total of 61 participants completed the final month 3 visit. The 11 participants lost to follow-up were treated as smokers for the purposes of data analysis.
Measure: Number; unit: participants
Arm/Group | Chantix for 3 Months, Standard Counseling | Chantix for 3 Months and Adherence Counseling
Number analyzed (Participants) | 36 | 36
participants | 9 (.422) | 8 (.439)

3. Secondary Outcome: Carbon Monoxide-verified Abstinence
Description: Carbon monoxide-verified abstinence determined as a measure of <10 ppm (parts per million). Less than 2ppm CO found in healthy non-smokers.
Time Frame: Month 1
Population: A total of 60 participants completed the month 1 visit. The 12 participants lost to follow-up were treated as smokers for the purposes of data analysis.
Measure: Number; unit: participants
Arm/Group | Chantix for 3 Months, Standard Counseling | Chantix for 3 Months and Adherence Counseling
Number analyzed (Participants) | 36 | 36
participants | 7 (.441) | 6 (.397)

4. Secondary Outcome: Carbon Monoxide-verified Abstinence
Description: as for outcome 3
Time Frame: Month 2
Population: A total of 57 participants completed the month 2 visit. The 15 participants lost to follow-up were treated as smokers for the purposes of data analysis.
Measure: Number; unit: participants
Arm/Group | Chantix for 3 Months, Standard Counseling | Chantix for 3 Months and Adherence Counseling
Number analyzed (Participants) | 36 | 36
participants | 6 (16.981) | 5 (18.931)

ADVERSE EVENTS:
Arm/Group | Chantix for 3 Months, Standard Counseling | Chantix for 3 Months and Adherence Counseling
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36
Other Adverse Events (participants affected / at risk) | 12/36 | 14/36
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chantix for 3 Months, Standard Counseling (N=36) | Chantix for 3 Months and Adherence Counseling (N=36)
Nausea (Gastrointestinal disorders) | 9 | 9
Gas (Gastrointestinal disorders) | 12 | 12
Dry Mouth (Gastrointestinal disorders) | 7 | 12
Headaches (General disorders) | 7 | 13
constipation (General disorders) | 4 | 8
Trouble sleeping (General disorders) | 9 | 14
Irritability (General disorders) | 6 | 13
Dizziness (General disorders) | 4 | 6
Fatigue (General disorders) | 10 | 9
Abnormal Dreams (General disorders) | 6 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes